CLINICAL TRIAL: NCT06781671
Title: Supportive Nursing Care for İCU Patients, Structured According to Comfort Theory
Brief Title: Use of Comfort Theory In Intensive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SAÜ-SBE-FK-01
Record Dates: First submitted 2024-01-21; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Intensive Care Unit
Keywords: Comfort Theory; Nursing Care; Video Interview; Radio-Television; Environmental Stress

STUDY DESIGN:
Intervention Model Description: The groups will be divided into two based on hospital protocol numbers. Those with an even protocol number will be included in the intervention group, while those with an odd number will be included in the control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in the control group were subjected to standard intensive care conditions Routine monitoring and treatments were administered. Repositioning was performed for patients in need every two hours within the bed Visits were conducted daily with a maximum duration of five minutes per patient, allowing only one family member to be present face-to-face.
  Each night at 01:00, a routine chest X-ray was taken*, and routine blood samples** were collected at 03:00.
  Mobilization was not carried out during the day unless deemed necessary. Patients did not receive any materials such as tablet computers, sleep masks, or sleep headphones The Patient Identification Form, General Comfort Scale, and Intensive Care Unit Environmental Stressor Scale were administered face-to-face by the researcher 48 hours after the patient admission to the intensive care unit.
  = Since the researched department is the intensive care unit for chest diseases, routine chest X-rays are taken from patients every nigt
- Intervention (Experimental): Structured nursing interventions based on the Comfort Theory were applied to patients in the intervention group. Patients were mobilized at least once during the day. Auxiliary materials believed to increase patient comfort, such as tablet computers, wired headphones, sleep headphones, and sleep masks, were provided. Patients had face-to-face meetings with their families during the day and video calls in the evening. Care interventions were minimized as much as possible for patients between 24:00-07:00 at night, and treatments were carefully planned around these hours. Blood sampling was performed at 23:00 at night, and X-rays were taken at 07:00 in the morning. The Patient Identification Form, General Comfort Scale, and Intensive Care Unit Environmental Stressor Scale were administered face-to-face by the researcher 48 hours after the patient&#39;s admission to the intensive care unit.
  Interventions: Behavioral: ComfortTheory

INTERVENTIONS:
Behavioral: ComfortTheory — Structured nursing interventions based on the Comfort Theory were applied to patients in the intervention group.
  Patients were mobilized at least once during the day. Auxiliary materials believed to increase patient comfort, such as tablet computers, wired headphones, sleep headphones, and sleep masks, were provided.
  Patients had face-to-face meetings with their families during the day and video calls in the evening.
  Care interventions were minimized as much as possible for patients between 24:00-07:00 at night, and treatments were carefully planned around these hours.
  Blood sampling was performed at 23:00 at night, and X-rays were taken at 07:00 in the morning.
  The Patient Identification Form, General Comfort Scale, and Intensive Care Unit Environmental Stressor Scale were administered face-to-face by the researcher 48 hours after the patient&#39;s admission to the intensive care unit.
  Other Names: Intervention Group
  Arms: Intervention

SUMMARY:
Nursing interventions, which has been configured to conform In this study, the mutual comfort needs of intensive care patients that were supported by various materials such as tablet computers and remote video call systems ,which was configured according to the comfort theory and applied to patients in the form of nursing interventions.. It was planned to examine that the effects of nursing interventions which was structured according to the comfort theory, applied to patients on the comfort levels of the patients and their perceived environmental stressor levels.

DETAILED DESCRIPTION:
1.1 PROBLEM DEFINITION AND IMPORTANCE

Intensive care units (ICUs) are specialized units where critical care is provided to patients with life-threatening conditions, requiring life-supporting treatment and continuous monitoring. These units operate in intense and stressful environments, utilizing specialized and advanced treatment methods with a multidisciplinary team approach, alongside complex biomedical devices. Patients in the ICU are confined to a limited environment, connected to equipment for treatment and monitoring 24 hours a day. They are exposed to physical factors such as noise, light, room temperature fluctuations, and frequent care and treatment activities. Additionally, patients in the ICU experience emotional challenges and high levels of stress, including being away from their families, witnessing treatments and interventions on other patients, and dependence on healthcare providers for treatment and care. All these complex processes adversely affect the comfort of patients in physical, sociocultural, psychospiritual, and environmental dimensions.

A healthy ICU should be designed to motivate the patient's participation in treatment and care, aiming to facilitate recovery. Improving patient comfort in the intensive care unit will enhance the quality of nursing care and shorten the recovery period. Various models and theories exist to enhance and standardize the quality of nursing care with the aim of increasing patient comfort. The Comfort Theory, developed by Kolcaba and based on the nursing function of relief, forms the foundation for nursing care. Kolcaba spent 15 years developing the concept of comfort and its application to patient comfort, creating a taxonomic structure consisting of three levels and four dimensions in 1988. Kolcaba described the concept of comfort, explained holistically, as the current experience of meeting basic human needs for relief, ease, and overcoming problems.

Studies in the literature indicate that high-quality nursing care based on the Comfort Theory positively influences comfort. Patients often report factors that disrupt their comfort after discharge from the ICU and lead to distress, such as sleep-related problems, pain, dehydration, orientation or consciousness disorders, anxiety, loss of appetite, noise, weakness, inability to communicate with the environment, and endotracheal tube application. Conversely, factors that enhance their comfort and make them feel good include feeling safe and the presence of nurses. The main negative environmental features of ICUs reported by patients include high noise levels, artificial lighting, an unfamiliar environment, the presence of complex devices, and the absence of devices such as TV and radio, which reduce comfort. These negative environmental features of ICUs decrease patient comfort and increase the level of stress they experience. Moreover, stressors in the ICU lead to sensory overload, perceptual deprivation, and the development of intensive care syndrome. Stress and related disorders experienced by patients in the ICU have a negative impact on individuals' health, prolong the healing process, and increase the length of hospital stays.

When reviewing studies that base nursing care on the Comfort Theory in the literature, it is observed that these studies are conducted in various fields of nursing, such as perianesthesia, urogynecology, oncology, cardiology, psychiatry, and end-of-life care. Interventions based on this theory have been found to positively affect patients' comfort. In Turkey, however, there is limited research on nursing practices based on the Comfort Theory. In a study conducted by Karabacak (2004) with breast cancer patients, it was reported that comfort-supportive nursing care reduced anxiety and increased adherence to radiotherapy. In a study conducted by Yeşim and Türkan (2017), nursing care based on the Comfort Theory in the postpartum period was found to increase the comfort levels of women undergoing cesarean section. Zengin (2012), in his study, emphasized that nursing interventions based on the Comfort Theory, supported by the literature, could be effective in intensive care patients.

Considering the comfort and stress levels of ICU patients, it is necessary to improve and update nursing care, create alternative care methods, and make them applicable to ICU patients. In light of this information, when observations in the ICU and literature information are compiled, it is believed that nursing care structured according to the Comfort Theory will have positive contributions to ICU patients, enhance the quality of care, and guide the development of similar nursing interventions.

1.2 OBJECTIVE OF THE RESEARCH

This study is designed to examine the impact of structured supportive nursing care for intensive care unit (ICU) patients on the environmental stressors perceived by patients in the ICU and on the fundamental factors influencing patients' comfort at a basic level, including physical, environmental, sociocultural, and psychospiritual factors (such as separation from normal life, restricted communication with family/relatives, and inappropriate environmental conditions).

METHODOLOGY

The study, designed with an experimental design comprising a control group (n:25) and an intervention group (n:25), was planned in accordance with a randomized controlled research design. Initially, the common comfort needs of intensive care unit (ICU) patients were identified, and nursing care plans structured according to the Comfort Theory for ICU patients were created. While patients in the control group were monitored under standard ICU conditions, structured nursing interventions will be applied to patients in the intervention group. The data of the study will be collected using the Patient Identification Form; General Comfort Scale and Intensive Care Unit Environmental Stressor Scale; Parametric tests will be utilized in the evaluation of study data.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old or older
* Requiring intensive care treatment for at least 48 hours
* Being literate
* Having no sensory losses such as vision, hearing, or speech impairments
* Being open to communication and collaboration
* Currently undergoing treatment in the intensive care unit
* Approval from both the patient and the family to participate in the study
* Sufficient knowledge on the part of the patient's family for remote video communication

Exclusion Criteria:

* Not meeting the inclusion criteria
* Refusing consent at any stage of the study and withdrawing from the study
* Being intubated
* Having cognitive disorders such as dementia, Alzheimer's, and Parkinson's
* Discharged from the intensive care unit before 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Are supportive nursing care interventions structured according to Kolcaba's Comfort Theory more effective than standard nursing care in increasing patients' comfort levels? | Minimum 48 hours
  Supportive nursing care structured according to the comfort theory applied to intensive care patients for 48 hours increased the comfort level of patients.
  General Comfort Scale: The Turkish validity and reliability study of the General Comfort Scale developed by Katharine Kolcaba in 1992 was conducted by Kuguoglu and Karabacak. The scale is a four-point Likert-type and consists of 48 items. The comfort levels of the scale are relief (16 items), relaxation (17 items) and superiority (15 items). The scale consists of positive and negative items and these items are mixed. The highest total score that can be obtained from the scale is 192, while the lowest total score is 48. Low comfort is expressed with one point and high comfort is expressed with four points. In the validity and reliability study, the Cronbach alpha coefficient of the scale was found to be 0.85. For this study group, the Cronbach alpha coefficient of the scale was found to be 0.91.

SECONDARY OUTCOMES:
Are supportive nursing care interventions structured according to Kolcaba's Comfort Theory effective in reducing environmental stress compared to standard nursing care? | Minimum 48 hours
  Supportive nursing care structured according to the comfort theory applied to intensive care patients for 48 hours reduced the level of stress perceived by patients in intensive care.
  Intensive Care Environmental Stressor Scale: It was developed by Ballard in 1981 to describe the stressors perceived by patients treated in the intensive care unit and was revised by Cochran and Ganong in 1989. The scale was adapted into Turkish by Aslan (2010) and Cronbach's alpha coefficient was found to be 0.94. The four-point Likert-type scale consists of 42 items. The highest total score that can be obtained from the scale is 168 and the lowest total score is 42. The high score obtained from the scale indicates that environmental stressors perceived in intensive care negatively affect patients.For this study group, the Cronbach alpha coefficient of the scale was found to be 0.94

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya Universty, Sakarya, Serdivan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No